CLINICAL TRIAL: NCT06457308
Title: Tainan Hospital, Ministry of Health and Welfare, Taiwan
Brief Title: Compare the Agility Exercise and Resistance Exercise on Physical Function and Stability in Osteoporotic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tainan Hospital, Ministry of Health and Welfare (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TainanHMHW
Record Dates: First submitted 2024-04-06; First posted 2024-06-13 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Postmenopausal Osteoporosis; Agility Exercise; Physical Function; Balance Stability; Fall Prevention
Keywords: postmenopausal osteoporosis; agility exercise; physical function; multi-component exercise; fall prevention
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Intervention Model Description: Non-randomized, quasi-experimental design.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Agility exercise training. (Experimental): Participants attend training class focused on agility training. Rope ladders and cones are used to perform multiple tasks of direction changes, acceleration and deceleration of footsteps, hand and foot coordination and spatial orientation training.
  Interventions: Biological: Physical training of agility
- Resistance exercise training. (Active Comparator): Participants attend training class focused on resistance training. Resistance training for upper and lower limb muscles and core muscles, including squats, use of elastic bands, and simple bars.
  Interventions: Biological: Physical training of resistance
- Control (No Intervention): Participants only receive osteoporosis education usual care.

INTERVENTIONS:
Biological: Physical training of agility — A grouped training for older adults in the community. The training classed lasted for 12 weeks, one session a week for 120 mins, and are under instructed by a trained experienced sport instructor. Use rope ladders and cones to perform multiple tasks of direction changes, acceleration and deceleration of footsteps, hand and foot coordination and spatial orientation training,
  Arms: Agility exercise training.
Biological: Physical training of resistance — A grouped training for older adults in the community. The training classed lasted for 12 weeks, one session a week for 120 mins, and are under instructed by a trained experienced sport instructor. Resistance training for upper and lower limb muscles and core muscles, including squats, use of elastic bands, and simple bars
  Arms: Resistance exercise training.

SUMMARY:
Osteoporosis weakens bones with age, increasing fracture risk. Exercise improves physical function and reduces falls, crucial for preventing osteoporotic fractures, especially with balance, resistance, and multi-component training. Agility exercise, integrating various aspects like aerobic, strength, balance, and cognitive tasks, is promising for fall prevention in older adults, though its effectiveness in osteoporosis is not extensively studied.

This study compares agility and resistance exercise impacts on physical function and balance stability in postmenopausal osteoporosis. Fifty-one women (average age: 68±6.3y, BMI: 22.3±2.7 kg/m2) were divided into agility exercise (AG), resistance exercise (RG), and control groups (CG) through purposive sampling. AG and RG received added intervention training once a week for 2 hours over 12 weeks. Main outcomes included physical function and balance stability measured through various tests.

DETAILED DESCRIPTION:
Main activities of agility training group (AG): Use rope ladders and cones to perform multiple tasks of direction changes, acceleration and deceleration of footsteps, hand and foot coordination and spatial orientation training.

Main activities of resistance training group (AG): Resistance training for upper and lower limb muscles and core muscles, including squats, use of elastic bands, and simple bars.

ELIGIBILITY:
Inclusion Criteria:

* women with osteoporosis( diagnosed with DXA, T-score≦-2.5 in L-spine or hip)
* postmenopausal, more than 50 years old,

Exclusion Criteria:

* unable to attend the training sessions due to physical problems
* had joined previous exercise program

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — postmenopausal osteoporosis
Enrollment: 51 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Physical function of upper limb strength | after the completed training course, about 12 weeks
  arm curl in 30 secs
Physical function of upper limbs strength | after the completed training course, about 12 weeks
  Hand grip
Physical function of lower limbs | after the completed training course, about 12 weeks
  Walking speed
Physical function of dynamic balance | after the completed training course, about 12 weeks
  Up and go test
Physical function of lower limbs | after the completed training course, about 12 weeks
  Sit to stand in 30 secs
Physical function of static balance | after the completed training course, about 12 weeks
  One leg stand test
Stability index | after the completed training course, about 12 weeks
  Biodex balance system device

CONTACTS AND LOCATIONS:
Locations (1):
- Chen, Ying-Chen, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donath L, van Dieen J, Faude O. Exercise-Based Fall Prevention in the Elderly: What About Agility? Sports Med. 2016 Feb;46(2):143-9. doi: 10.1007/s40279-015-0389-5. PMID 26395115
- [Background] Lichtenstein E, Morat M, Roth R, Donath L, Faude O. Agility-based exercise training compared to traditional strength and balance training in older adults: a pilot randomized trial. PeerJ. 2020 Apr 14;8:e8781. doi: 10.7717/peerj.8781. eCollection 2020. PMID 32328344
- [Background] Morat M, Morat T, Zijlstra W, Donath L. Effects of multimodal agility-like exercise training compared to inactive controls and alternative training on physical performance in older adults: a systematic review and meta-analysis. Eur Rev Aging Phys Act. 2021 Feb 25;18(1):4. doi: 10.1186/s11556-021-00256-y. PMID 33632117
- [Background] Miko I, Szerb I, Szerb A, Bender T, Poor G. Effect of a balance-training programme on postural balance, aerobic capacity and frequency of falls in women with osteoporosis: A randomized controlled trial. J Rehabil Med. 2018 Jun 15;50(6):542-547. doi: 10.2340/16501977-2349. PMID 29767227